CLINICAL TRIAL: NCT02226406
Title: Effect of Early Physical Exercise on Pulmonary Ventilation and Recruitment Evaluated With Electric Impedance Tomography.
Brief Title: Effect of Early Physical Exercise on Pulmonary Ventilation and Recruitment
Acronym: EFRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EIT-Early Exercise
Record Dates: First submitted 2014-07-31; First posted 2014-08-27 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Critical Illness
Keywords: Early Physical Exercise; Alveolar Recruitment; Electrical Impedance Tomography; Oxygenation; Ventilation
MeSH Terms: conditions — Critical Illness; Motor Activity; Respiratory Aspiration | interventions — Early Ambulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Legs Cycloergometer Group (A) (Experimental): Patients randomized in this group will do 10 minutes of legs cycloergometer active exercise. Continuously evaluated with electric impedance tomography.
  Interventions: Other: A: Chair - Leg Cycle ergometer
- Hands Cycloergometer Group (B) (Experimental): Patients randomized in this group will do 10 minutes of hand cycloergometer active exercise. Continuously evaluated with electric impedance tomography.
  Interventions: Other: B: Chair - Arm Cycle ergometer
- Walk in place (C) (Experimental): Patients randomized in this group will do 10 minutes of active walk in place. Continuously evaluated with electric impedance tomography.
  Interventions: Other: C: Walk in place

INTERVENTIONS:
Other: A: Chair - Leg Cycle ergometer
  Other Names: Exercise Bike; Early mobilization; Early physical therapy; Early physical rehabilitation; Early physical training; Early physiotherapy; Very early mobilization; Early exercise; Early activity; Early mobility therapy
  Arms: Legs Cycloergometer Group (A)
Other: B: Chair - Arm Cycle ergometer
  Other Names: Handcycle; Early mobilization; Early physical therapy; Early physical rehabilitation; Early physical training; Early physiotherapy; Very early mobilization; Early exercise; Early activity; Early mobility therapy
  Arms: Hands Cycloergometer Group (B)
Other: C: Walk in place
  Other Names: Early mobilization; March; Static walk; Early physical therapy; Early physical rehabilitation; Early physical training; Early physiotherapy; Very early mobilization; Early exercise; Early activity; Early mobility therapy
  Arms: Walk in place (C)

SUMMARY:
In the critically patient bed rest and immobilization are some of the responsable of the development of respiratory complications. Early physical exercise is a tool to prevent respiratory complications as lost of respiratory muscle strength, decrease in functional residual capacity and hypoxemia improving oxygenation.

New technology as electrical impedance tomography (EIT) are available to visualize changes of regional lung aeration.

The aim of this study is to assess the effect of early physical exercise improving alveolar recruitment and pulmonary ventilation in intensive care unit (ICU) patients, evaluated with EIT.

The ICU patients included at day of evaluation will be evaluated continuously with EIT in different positions. 1) in the supine position (at 30° of inclination), 2) Sitting in chair 3) Active physical exercise 4) And rest in chair after exercise

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted at the Intensive Care Medical/Surgical Unit of Clinic Saint Luc
* Days of hospitalization between 1 and 10
* Hemodynamically stable
* Patient or family member sign the informed consent

Exclusion Criteria:

* With risk of evisceration
* Therapy withdrawal
* With cardiac devices (Pace Maker)
* Persistent cough
* Patches or open wounds in zone of electrodes
* Presence of high vasopressor medication (noradrenaline > 3 mg/h)
* PEEP > 15 cm H2
* Acute Myocardial Infarction
* Active bleeding
* Intracranial pressure > 20 mm Hg or with major instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in pulmonary electric impedance tomography (EIT) before, during and after single session of exercise. | Meassure of EIT after 10 minutes of exercise and will be compared with baseline EIT
  The change in pulmonary recruitment and ventilation will be evaluated with electric impedance tomography (EIT) in single session of exercise. First measure will be made for five minutes with EIT, before the exercise, then second measure will be made during exercise for ten minutes with EIT and finally last measure will be made after exercise for twenty minutes with EIT. All impedanciometries obtained in the patient in different activities will compare each.

SECONDARY OUTCOMES:
Change in PaO2 before, during and after single session of exercise | Measure of PaO2 after 20 minutes of exercise and will compared with baseline PaO2
  Before exercise will be taken a sample of arterial blood gases for determinate the initial PaO2 of the patient. Twenty minutes after exercise will be taken a new sample of arterial blood gases to establish the difference between PaO2 before exercise and after exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Arriagada, PT, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc); Ursula Jeria, PT, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc); Cheryl Hickmann, PT, PhD student, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc); Jean Roeseler, PT, PhD, Study Director — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc); Pierre-François Laterre, MD, Study Chair — Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc)
Locations (1):
- Cliniques universitaires Saint-Luc- Université Catholique de Louvain (StLuc), Brussels, Belgium